CLINICAL TRIAL: NCT01435655
Title: The Effect On Transthyretin Stabilization, Safety, Tolerablity, Efficacy And Pharmacokinetics Of Orally Administered Tafamidis In Transthyretin Amyloid Polyneuropathy Patients With V30m Or Non-v30m Transthyretin: A Phase Iii, Open-label Study
Brief Title: The Effect Of Tafamidis For The Transthyretin Amyloid Polyneuropathy Patients With V30M Or Non-V30M Transthyretin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B3461010
Record Dates: First submitted 2011-09-13; First posted 2011-09-16 (Estimated); Results first posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-08

CONDITIONS: Transthyretin Familial Amyloid Polyneuropathy
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open (Experimental): tafamidis
  Interventions: Drug: tafamidis

INTERVENTIONS:
Drug: tafamidis — tafamidis meglumine 20 mg QD
  Other Names: tafamidis meglumine

SUMMARY:
Tafamidis has been developed as an oral specific stabilizer of transthyretin tetramer.

ELIGIBILITY:
Inclusion Criteria:

* Transthyretin amyloid polyneuropathy with V30M or non-V30M transthyretin mutation.
* Subject had amyloid documented by biopsy in accordance with institutional site standard of care.

Exclusion Criteria:

* Primary amyloidosis and secondary amyloidosis.
* History of liver transplant.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Japan (2):
  - Kumamoto University Hospital/Department of Neurology, Kumamoto, Kumamoto
  - Shinshu University Hospital/Department of Medicine (Neurology and Reumatology), Matsumoto-shi, Nagano

REFERENCES:
- [Derived] Huber P, Flynn A, Sultan MB, Li H, Rill D, Ebede B, Gundapaneni B, Schwartz JH. A comprehensive safety profile of tafamidis in patients with transthyretin amyloid polyneuropathy. Amyloid. 2019 Dec;26(4):203-209. doi: 10.1080/13506129.2019.1643714. Epub 2019 Jul 27. PMID 31353964
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461010&StudyName=The%20Effect%20Of%20Tafamidis%20For%20The%20Transthyretin%20Amyloid%20Polyneuropathy%20Patients%20With%20V30M%20Or%20Non-V30M%20Transthyretin

RESULTS

PARTICIPANT FLOW:
Groups:
- Tafamidis 20 mg: Participants (V30m and non-V30m transthyretin mutation) received tafamidis 20 mg soft gelatin capsules orally once daily for up to 78 weeks
Period: Overall Study
Arm/Group | Tafamidis 20 mg
Started | 10
Completed | 7
Not Completed | 3
Not completed — Death | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Transthyretin (TTR) Stabilization at Week 8 Compared With Baseline as Measured by a Validated Immunoturbidimetric Assay
Description: TTR tetramer level for each plasma sample was assessed using a validated immunoturbidimetric assay before and after urea denaturation. The Fraction of Initial (FOI) tetramer concentration is the ratio of the measured TTR tetramer concentration after denaturation to the measured TTR tetramer average concentration before denaturation. TTR tetramer stabilization is based on the difference between the on-treatment FOI and the baseline FOI expressed as a percentage of the baseline FOI. A patient who has the "TTR stabilization" is defined as the patient whose percent stabilization is equal to or more than 32%.
Time Frame: 8 weeks
Population: Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS); NIS (Total), NIS-LL (Lower Limb) and NIS-UL (Upper Limb) at Week 26, Week 52 and Week 78
Description: The NIS provides a total body single score of neuropathic deficits (score range: 0-122, higher score = more deficit), comprising subset scores for cranial nerves, muscle weakness, reflexes, and sensation (based on mean of 2 scores in 1 week period; each item scored separately for left and right). The NIS-LL is a subscale that provides a score for the lower limbs functions (muscle weakness, reflexes and sensation in great toe) and has a score range of 0-44 (higher score = more deficit). The NIS-UL is a subscale that provides a score for the upper body functions (muscle weakness [including cranial nerves], reflexes and sensation in finger) and has a score range of 0-78 (higher score = more deficit). The components for cranial nerves and muscle weakness are scored from 0 (Normal) to 4 (Paralysis), and those for reflexes and sensation from 0 (Normal) to 2 (Absent). For all items, higher scores indicate greater impairment.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
Units on a scale
  NIS-Total: Baseline (n=10) | 31.03 (26.260)
  NIS-Total: Change at Week 26 (n=10) | 4.37 (9.408)
  NIS-Total: Change at Week 52 (n=10) | 8.30 (8.326)
  NIS-Total: Change at Week 78 (n=8) | 9.90 (12.584)
  NIS-LL: Baseline (n=10) | 16.99 (13.143)
  NIS-LL: Change at Week 26 (n=10) | 2.06 (5.565)
  NIS-LL: Change at Week 52 (n=10) | 3.62 (4.374)
  NIS-LL: Change at Week 78 (n=8) | 3.30 (4.739)
  NIS-UL: Baseline (n=10) | 14.03 (13.716)
  NIS-UL: Change at Week 26 (n=10) | 2.31 (4.066)
  NIS-UL: Change at Week 52 (n=10) | 4.68 (5.103)
  NIS-UL: Change at Week 78 (n=8) | 6.59 (8.724)

3. Secondary Outcome: Change From Baseline in Scores of the Total Quality of Life (TQOL) and 5 Domains as Measured by the Norfolk QOL - Diabetic Neuropathy (Norfolk QOL-DN) at Week 26, Week 52 and Week 78.
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire. It consists of 5 domains: Physical Functioning/Large Fiber [score range: -4 - 56] , Activities of Daily Living (ADL) [0 - 20], Symptoms [0 - 32], Small Fiber [0 - 16] and Autonomic [0 - 12]. Total of quality of life (TQOL) score is the sum of all five domains with a range of -4 to 136 (Pfizer Data Standards). Higher scores on each item of the Norfolk QOL-DN TQOL indicate worse quality of life.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
Units on a scale
  TQOL: Baseline (n=10) | 52.9 (32.76)
  TQOL: Change at Week 26 (n=10) | 11.8 (20.01)
  TQOL: Change at Week 52 (n=10) | 9.1 (12.49)
  TQOL: Change at Week 78 (n=8) | 10.8 (13.69)
  Physical Functioning: Baseline (n=10) | 25.6 (15.28)
  Physical Functioning: Change at Week 26 (n=10) | 4.8 (10.02)
  Physical Functioning: Change at Week 52 (n=10) | 2.2 (8.87)
  Physical Functioning: Change at Week 78 (n=8) | 4.1 (7.83)
  ADL: Baseline (n=10) | 8.5 (7.63)
  ADL: Change at Week 26 (n=10) | 1.2 (3.61)
  ADL: Change at Week 52 (n=10) | 0.8 (3.52)
  ADL: Change at Week 78 (n=8) | 0.6 (2.33)
  Symptoms: Baseline (n=10) | 8.5 (5.34)
  Symptoms: Change at Week 26 (n=10) | 2.6 (3.47)
  Symptoms: Change at Week 52 (n=10) | 4.0 (5.73)
  Symptoms: Change at Week 78 (n=8) | 3.1 (3.94)
  Small Fiber: Baseline (n=10) | 6.3 (5.31)
  Small Fiber: Change at Week 26 (n=10) | 1.9 (4.25)
  Small Fiber: Change at Week 52 (n=10) | 1.6 (2.32)
  Small Fiber: Change at Week 78 (n=8) | 2.1 (3.76)
  Autonomic: Baseline (n=10) | 4.0 (3.06)
  Autonomic: Change at Week 26 (n=10) | 1.3 (1.42)
  Autonomic: Change at Week 52 (n=10) | 0.5 (1.43)
  Autonomic: Change at Week 78 (n=8) | 0.8 (1.91)

4. Secondary Outcome: Change From Baseline in Summated 7 Nerve Tests Normal Deviate Score (∑ 7 NTs Nds) as Measured by Nerve Conduction Studies (NCS), Vibration Detection Threshold (VDT) and Heart Rate Response to Deep Breathing (HRDB) at Week 26, Week 52, and Week 78
Description: The Σ7 NTs nds measures primarily large-fiber function. It is a composite score derived from five NCS attributes (peroneal nerve distal motor latency, peroneal nerve compound muscle action potential, peroneal nerve motor conduction velocity, tibial nerve distal motor latency, and sural nerve sensory nerve action potential amplitude) along with VDT obtained in great toes by Quantitative Sensory Testing (QST), and HRDB value. It is defined as 7 times the mean of non-missing values of, the five normal deviates of NCS, HRDB, and average normal deviate for VDT of toes. Score was determined through reference to normal values for age, sex, height and abnormalities scored. Total score range is approximately -26 to 26, where higher score=worse nerve function.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
Units on a scale
  Baseline (n=10) | 8.33 (5.574)
  Change at Week 26 (n=10) | 0.55 (2.657)
  Change at Week 52 (n-=10) | 1.04 (2.992)
  Change at Week 78 (n=8) | 1.92 (5.129)

5. Secondary Outcome: Change From Baseline in Summated 3 Nerve Tests Small Fiber Normal Deviate Score (∑ 3 NTSF Nds) as Measured by Cooling and Heat Pain Thresholds by QST and HRDB at Week 26, Week 52 and Week 78
Description: The Σ3 NTSF nds measures small-fiber function. It is a composite score defined as 3 times the mean of non-missing values of normal deviates of cooling threshold for lower limbs, heat pain intermediate response for lower limbs, and HRDB. The total score range is approximately -11.2 to 11.2, with a higher score demonstrating worse nerve function.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
Units on a scale
  Baseline (n=10) | 6.39 (3.160)
  Change at Week 26 (n=10) | 0.16 (1.619)
  Change at Week 52 (n=10) | -0.13 (1.334)
  Change at Week 78 (n=8) | 0.40 (1.985)

6. Secondary Outcome: Change From Baseline in Modified Body Mass Index (mBMI) at Week 8, Week 26, Week 52 and End of Study
Description: The mBMI was calculated by multiplying the BMI (the weight in kilograms divided by the square of the height in meters) by serum albumin level (gram/liter). Change in mBMI was calculated as the mBMI at the given week minus the Baseline mBMI.
Time Frame: Baseline, Week 8, Week 26, Week 52, End of Study
Population: Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: (kilogram/square meter)*(gram/liter)
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
(kilogram/square meter)*(gram/liter)
  Baseline (n=10) | 805.70 (193.378)
  Change at Week 8 (n=10) | 74.86 (88.706)
  Change at Week 26 (n=10) | 26.61 (61.862)
  Change at Week 52 (n=10) | 64.86 (80.016)
  End of Study (n=7) | 53.65 (81.386)

7. Secondary Outcome: Change From Baseline in Ambulatory Status at Week 26, Week 52 and Week 78
Description: Ambulatory status was evaluated using walking ability scale in polyneuropathy disability score. The ambulatory status was evaluated as: 0=Good, 1=Sensory disturbances in the feet but able to walk without difficulty, 2=Some difficulties with walking but can walk without aid, 3a=Able to walk with 1 stick or crutch, 3b=Able to walk with 2 sticks or crutches, 4=Not ambulatory, confined to a wheelchair or bedridden.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
Participants
  Baseline (n=10): Status 0 | 0
  Baseline (n=10): Status 1 | 3
  Baseline (n=10): Status 2 | 4
  Baseline (n=10): Status 3a | 2
  Baseline (n=10): Status 3b | 1
  Baseline (n=10): Status 4 | 0
  Week 26 (n=10): Status 0 | 1
  Week 26 (n=10): Status 1 | 2
  Week 26 (n=10): Status 2 | 3
  Week 26 (n=10): Status 3a | 2
  Week 26 (n=10): Status 3b | 2
  Week 26 (n=10): Status 4 | 0
  Week 52 (n=10): Status 0 | 1
  Week 52 (n=10): Status 1 | 1
  Week 52 (n=10): Status 2 | 4
  Week 52 (n=10): Status 3a | 2
  Week 52 (n=10): Status 3b | 2
  Week 52 (n=10): Status 4 | 0
  Week 78 (n=8): Status 0 | 1
  Week 78 (n=8): Status 1 | 1
  Week 78 (n=8): Status 2 | 2
  Week 78 (n=8): Status 3a | 2
  Week 78 (n=8): Status 3b | 2
  Week 78 (n=8): Status 4 | 0

8. Secondary Outcome: Number of Participants With Transthyretin (TTR) Stabilization at Week 26, Week 52, and Week 78 Compared With Baseline as Measured by a Validated Immunoturbidimetric Assay
Description: TTR tetramer was assessed using a validated immunoturbidimetric assay. The TTR tetramer level for each plasma sample was measured before and after urea denaturation. The Fraction of Initial (FOI) tetramer concentration is the ratio of the measured TTR tetramer concentration after denaturation to the measured TTR tetramer concentration before denaturation. TTR tetramer stabilization is based on the difference between the on-treatment FOI and the baseline FOI expressed as a percentage of the baseline FOI. A patient who has the "TTR stabilization" is defined as the patient whose percent stabilization is equal to or more than 32%.
Time Frame: Baseline, Week 26, Week 52, Week 78
Population: Full Analysis Set (FAS) included all participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
Participants
  Week 26 | 10
  Week 52 | 9
  Week 78 | 8

9. Other Pre Specified Outcome: Plasma Concentration of Tafamidis at Week 8, Week 26, Week 52 and Week 78
Description: Mean plasma concentration of tafamidis at 3 hours after administration
Time Frame: Week 8, Week 26, Week 52, Week 78
Population: The PK Analysis Set included all participants treated who had at least 1 quantifiable plasma tafamidis concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 10
ng/mL
  Week 8 (n=10) | 2773.0 (1777.71)
  Week 26 (n=10) | 2739.0 (1893.25)
  Week 52 (n=10) | 2829.0 (2315.58)
  Week 78 (n=8) | 3655.0 (2268.08)

ADVERSE EVENTS:
Arm/Group | Tafamidis 20 mg
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis 20 mg (N=10)
Atrioventricular block second degree (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Sudden death (General disorders) | 1
Pneumonia bacterial (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 1
Burns third degree (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Completed suicide (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis 20 mg (N=10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye discharge (Eye disorders) | 1
Vitreous opacities (Eye disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Paraesthesia oral (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Oral herpes (Infections and infestations) | 1
Tinea capitis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Gynaecomastia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.